CLINICAL TRIAL: NCT01321749
Title: The Neuroprotective Effect of Remote Ischemic Preconditioning on Ischemic Cerebral Vascular Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Ji Xunming, Xuan Wu Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RIPC2011
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Results first posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-03

CONDITIONS: Cerebrovascular Disease
Keywords: ischemic cerebral vascular disease; stroke secondary prevention; remote ischemic preconditioning
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIPC+stroke secondary prevension (Experimental): Procedure/Surgery: Remote Ischemic Preconditioning (RIPC) The detail of RIPC included five cycles of bilateral upper limbs 5/5 min. of ischemia and reperfusion alternation. Limb ischemia was induced by inflating tourniquets to 200 mmHg. This process was placed on both arms every day.
  Procedure:stroke secondary prevention(Such as Antiplatelet therapy, Cholesterol-lowering therapymaintain blood pressure and blood sugar normal)
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- stroke secondary prevention (No Intervention): Procedure:stroke secondary prevention(Such as Antiplatelet therapy, Cholesterol-lowering therapymaintain blood pressure and blood sugar normal)

INTERVENTIONS:
Procedure: Remote ischemic preconditioning (RIPC) — The detail of RIPC included five cycles of bilateral upper limbs 5/5 min. of ischemia and reperfusion alternation. Limb ischemia was induced by inflating tourniquets to 200 mmHg. This process was placed on both arms every day.
  Arms: RIPC+stroke secondary prevension

SUMMARY:
This study is a prospective, randomized, single-center trial, designed to observe the effect of remote limb ischemic preconditioning on ischemic cerebral vascular disease.

ELIGIBILITY:
Inclusion criteria:

1. Patients with stroke or transient ischemic attack (TIA) within 180 days and the neurologic deficits were well matched to the territory of the stenosed artery, with intracranial arterial stenosis of at least 50% by angiography, at least 70% by ultrasound, or at least 70% by computed tomographic angiography (CTA) or magnetic resonance angiography (MRA)
2. Age between 18 to 80 years old
3. Trial of Org 10172 in Acute Stroke Treatment-1 (TOAST-1) subtype
4. National Institutes of Health Stroke Scale (NIHSS) score 0-15, and Modified Rankin Scale (mRS) score 0-4.
5. ABCD2 score between 6 to 7
6. Stable vital signs, normal hepatic and renal functions,
7. No hemorrhagic tendencies.

Exclusion criteria:

1. Within 72 hrs of intra-artery or intravenous thrombolysis
2. Intracranial hemorrhage or large area of cerebral infarction (more than 1/3 middle cerebral artery perfusion territory)
3. Any soft tissue, orthopedic, or vascular injury, wounds or fractures in extremities which may pose a contraindication for application of the preconditioning cuffs
4. Acute myocardial infarction
5. Systolic blood pressure more than 200 mmHg after drug control
6. Peripheral blood vessel disease
7. Hematologic disease
8. Severe hepatic and renal dysfunction
9. Severe or unstable concomitant disease
10. Cannot tolerate BLIPC or without informed consent
11. Patients who did not complete the whole treatment procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Xicheng District, Beijing P.R., China

RESULTS

PARTICIPANT FLOW:
Groups:
- RIPC+Stroke Secondary Prevension: Procedure/Surgery: RIPC The detail of RIPC included five cycles of bilateral upper limbs 5/5 min. of ischemia and reperfusion alternation. Limb ischemia was induced by inflating tourniquets to 200 mmHg. This process was placed on both arms every day.
  Procedure:stroke secondary prevention
- Stroke Secondary Prevention: Procedure:stroke secondary prevention
Period: Overall Study
Arm/Group | RIPC+Stroke Secondary Prevension | Stroke Secondary Prevention
Started | 51 | 52
Completed | 38 | 30
Not Completed | 13 | 22
Not completed — Lost to Follow-up | 4 | 11
Not completed — Protocol Violation | 4 | 7
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RIPC+Stroke Secondary Prevension | Stroke Secondary Prevention | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 63
  >=65 years | 20 | 20 | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (10.1) | 60 (9.4) | 60.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  China | 51 | 52 | 103

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure and Heart Rates;
Time Frame: at the time points of baseline and 1, 15 and 30 days after BLIPC treatment
Reporting Status: Not Posted

2. Primary Outcome: Plasma Biomarkers of Coagulation and Fibrinolysis
Description: blood samples were collected one hour after every times of BLIPC procedure ended, and assayed with the immuno-turbidimetry assay on the coagulation laboratory autoanalyzer
Time Frame: the time points of baseline and 1, 15 and 30 days after BLIPC treatment
Reporting Status: Not Posted

3. Primary Outcome: Number of Patients Who Got New Brain Lesions
Description: We compared the number of patients who got new lesions in the Diffusion-weighted magnetic resonance imaging (DWI-MRI)
Time Frame: 300 days after treatment
Measure: Number; unit: participants
Arm/Group | RIPC+Stroke Secondary Prevension | Stroke Secondary Prevention
Number analyzed (Participants) | 38 | 30
participants | 3 | 8
Statistical Analysis 1: Comparison: RIPC+Stroke Secondary Prevension vs Stroke Secondary Prevention; Test type: Superiority or Other; p < 0.05, Log Rank

4. Secondary Outcome: The Time Point Until the First Stroke Recurrence,
Description: These patients underwent MRI/DWI at the time of first recurrence; patients without symptoms recurrence underwent follow-up MRI/DWI at 300 days.
Time Frame: At the 300-day after the initial treatment
Reporting Status: Not Posted

5. Secondary Outcome: Brain Perfusion Improvement Are Evaluated With SPECT and TCD
Description: Brain perfusion status were evalvated by SPECT SPECT scanning was performed using a dual headed rotating gamma camera at 30 minutes after intravenous 99mTc-ECD (25mCi) bolus injection and at 40 minutes after 18F -FDG bolus injection.
Time Frame: 300-day after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | RIPC+Stroke Secondary Prevension | Stroke Secondary Prevention
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 3/51 | 0/52
OTHER ADVERSE EVENTS (reported when occurring in more than 2.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIPC+Stroke Secondary Prevension (N=51) | Stroke Secondary Prevention (N=52)
transient sporadic subcutaneous bleeding points (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No